CLINICAL TRIAL: NCT04652401
Title: Assessment of Quality of Life and Its Determinants in Ventilator-dependent Patients With Slowly Progressive Neuromuscular Disease
Brief Title: Quality of Life in Ventilator-dependant Neuromuscular Patients
Acronym: EqualVENT
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other); AFM Téléthon (Unknown); FilNeMus (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A00997-32
Record Dates: First submitted 2020-11-09; First posted 2020-12-03 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Neuromuscular Diseases; Respiration, Artificial; Tracheostomy; Noninvasive Ventilation; Quality of Life
MeSH Terms: conditions — Neuromuscular Diseases; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at evaluating the quality of life of patients with slowly progressive neuromuscular disorders who are dependant on mechanical ventilation (daily usage ≥ 16h).

ELIGIBILITY:
Inclusion Criteria:

* Patients with slowly progressive neuromuscular disorder (NMD), non walking
* Patients dependant on mechanical ventilation (daily usage ≥ 16h) for at least 1 year before inclusion
* Aged ≥ 18 yo
* Consent for participation
* Affiliated to a social security regime

Exclusion Criteria:

* Patients with medically non-stable NMD: fever, acute respiratory infection, organ decompensation
* Patients with significant cognitive impairment (inability to read and/or incomprehension of questions)
* Patients with fast-evolving neuromuscular disease
* Patients declining to participate in the study
* Patients under guardianship and/or trusteeship
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with slowly progressive neuromuscular disease using home mechanical ventilation for at least 16 hours a day since at least one year. Patients may be ventilated via invasive or noninvasive interface.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Score of the Severe Respiratory Insufficiency questionnaire (SRI) | 1 Day
  Higher score represents better quality of life
Score of the Quality of Life Measure for people with slowly progressive and genetic neuromuscular disease questionnaire (QoL-gNMD) | 1 Day
  Higher score represents better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Delorme, MSc, Principal Investigator — Université Paris-Saclay, UVSQ, ERPHAN, 78000, Versailles, FRANCE; Frederic Lofaso, MD, PhD, Study Director — Université Paris-Saclay, UVSQ, ERPHAN, 78000, Versailles, FRANCE
Locations (1):
- AFM Téléthon, Évry, France

IPD SHARING:
Plan to Share IPD: No